CLINICAL TRIAL: NCT06811987
Title: Instructor-led Artificial Intelligence-Based Emergency Triage Education Tool in Enhancing Clinical Critical Thinking and Triage Practice: Randomized Control Trial
Brief Title: Artificial Intelligence-Based Emergency Triage Education Tool in Enhancing Clinical Critical Thinking and Triage Practice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HE-SF2024/57
Record Dates: First submitted 2025-01-16; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Nursing Teaching Pedagogy; Conversational AI Nursing Education Serious Game

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instructor-led (Active Comparator)
  Interventions: Behavioral: Instructor-led AI-Triage educational serious game
- Self-play (Experimental)
  Interventions: Behavioral: Self play AI-Triage educational serious game

INTERVENTIONS:
Behavioral: Instructor-led AI-Triage educational serious game — Participants will use the AI-triage serious game guided by the instructors.
  Arms: Instructor-led
Behavioral: Self play AI-Triage educational serious game — Participants will self-play the AI-Triage serious game during the class.
  Arms: Self-play

SUMMARY:
The study aims to develop an artificial intelligence (AI) based emergency triage education tool for providing critical thinking and questioning skills training to nursing students. It also aims to contribute valuable implications by collecting the knowledge, attitudes, and compassion aspects of nursing students toward AI-based education

The objectives of the study:

1. To evaluate the effectiveness of instructor-led and self-play pedagogy approaches in enhancing students' critical thinking by an AI-based emergency triage education tool.
2. To evaluate the effectiveness of instructor-led and self-play pedagogy approaches in enhancing students' triage skill retention by an AI-based emergency triage education tool.
3. To evaluate students' learning motivation, simulation-based experience, and usability towards AI-based technology learning.

Participants will

1. play the education tool in different pedagogy approaches
2. answer the questionnaires and receive a qualitative interview

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above;
2. Currently studying the NURS 225F of the Bachelor of Nursing (General) at Hong Kong Metropolitan University;
3. Able to use electronic devices to accomplish an online survey and participate in the AI-based emergency triage education tool

Exclusion Criteria:

* Currently working in emergency department

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-03-06 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Triage skill retention | Baseline, 1 month and 1 year
  short-term and long-term triage skill retention based on different pedagogy approaches The checklist is based on the Hospital Authority, Hong Kong triage guidelines. There are a total of 35 items that test the triage practice's specificity, which focuses on triage questioning and assessment selection in the game scenarios.
  For every corrected item, 1 score will be given. Therefore the maximum value is 35, presenting the best outcome in skill specificity; the minimum value is 0, the worst outcome.
  Moreover, 4 items are testing the triage accuracy of decision-making and management. The maximum value is 4, presenting the best outcome in skill accuracy; the minimum value is 0, the worst outcome.

SECONDARY OUTCOMES:
Cognitive Engagement | Immediately post intervention
  The cognitive engagement will be using the Situational Cognitive Engagement Measurements tools to evaluate.
  The tool consisted of three elements, measured by four items: (1) engagement with the task at hand, (2) effort and persistence, and (3) experience of flow or having been totally absorbed by the activity. The items were scored on a 5-point Likert scale: 1 (not true et al for me), 2 (not true for me), 3 (neutral), 4 (true for me), and 5 (very true for me). A higher total score presents a better cognitive engagement.
  Moreover, qualitative interviews to ask about their feeling and experiences towards cognitive engagement during the intervention.
Critical thinking | Base-line and 1 Month
  To evaluate the effectiveness of different pedagogies on students' critical thinking, the tool of Northeastern Illinois University's Critical Thinking Rubric is used to assess.
  Student performance is evaluated across four proficiency levels, ranging from 'limited or no proficiency' (scored at one point) to 'high proficiency' (scored at four points). The total rubric scores for a simulated scenario ranged from 6 to 24 (Higher scores represented a better critical thinking performance). is a comprehensive tool to assess critical thinking skills in six key dimensions.
Self-rated critical thinking | Baseline, 1 month
  by different pedagogies, the tool of Short Form English version of the Critical Thinking Disposition Inventory will be used to evaluate students' self-rated critical thinking index.
  It includes a series of statements related to critical thinking on a Likert scale (1: strongly disagree; 5: strongly agree), The tool may cover systematic analysis (5 items), thinking within the box (8 items) and outside the box (5 items). A higher score means better self-rated critical thinking.
Usability | Immediately post intervention
  The usability will be using the System Usability Scale tools to evaluate. The tool measured 10 items. The items were scored on a 5-point Likert scale: 1 (strongly disagree) to 5 (strongly agree). A higher total score presents a better system usability.
  Moreover, qualitative interviews to ask about their feeling and experiences towards system usability during the intervention.
simulation-based experience | Immediately post intervention
  The simulation-based experience will be using the Simulation Effectiveness Tool - Modified tools to evaluate.
  It is a 19-item tool that includes a 2-item pre-briefing, a 12-item scenario and a 5-item debriefing. A higher score on the tool reflects students' favourable perceptions of the simulation. Moreover, qualitative interviews to ask about their feeling and experiences towards simulation-based experience during the intervention.